CLINICAL TRIAL: NCT07044232
Title: NICardipine for Fast Achievement of Systolic BP Targets in ICH - a Quasi-randomized, Implementation Trial With Stepwise Rollout of Nicardipin Based Treatment of Hypertension.
Brief Title: NICardipine for Fast Achievement of Systolic BP Targets in ICH
Acronym: NICFAST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Rolf Blauenfeldt, MD, PhD, Associate Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NICFAST
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Intracerebral Haemorrhage
Keywords: Intracerebral Haemorrhage; blood pressure treatment; acute blood pressure treatment; nicardipine; glyceryl trinitrate
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Nicardipine; Labetalol; Methyldopa; Nitroglycerin; Nimodipine

STUDY DESIGN:
Intervention Model Description: Prospective, quasi-randomized, implementation and quality improvement trial with stepwise rollout
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors for 90 days modified Rankin Scale
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicardipine infusion based acute blood pressure lowering treatment (Experimental): 1. Nicardipine : Infusion at 5 mg/hour ( 2.5 mg/hour in renal or hepatic impairment and elderly. Taper after 4-6 hours.
  2. Labetalole: Dose: 10-20 mg IV, repeat as needed.
  3. Methyldopa: Dose: 250 mg three times daily (max 500 mg four times daily) orally or via feeding tube
  Acute antihypertensive treatment duration <72 hours
  Interventions: Combination Product: Nicardipine
- Glyceryl trinitrate patchbased acute blood pressure lowering treatment (Active Comparator): 1. Glyceryltrinitrate : Patch 5 or 10mg/24hour.
  2. Labetalole: Dose: 10-20 mg IV, repeat as needed.
  3. Nimotope: Dose: 30 or 60mg x 6 orally or via feeding tube
  Acute antihypertensive treatment duration <72 hours
  Interventions: Combination Product: Glyceryl trinitrate

INTERVENTIONS:
Combination Product: Nicardipine — Nicardipine infusion based acute blood pressure lowering treatment
  Other Names: Labetalol; Methyldopa
  Arms: Nicardipine infusion based acute blood pressure lowering treatment
Combination Product: Glyceryl trinitrate — Glyceryltrinitrate based acute blood pressure lowering treatment
  Other Names: Labetalol; Nimotop
  Arms: Glyceryl trinitrate patchbased acute blood pressure lowering treatment

SUMMARY:
Quality improvement study with a quasi-randomized design. The study monitors the effect of a gradually implemented treatment algorithm prioritizing intravenous antihypertensives (e.g., nicardipine) over long-acting nitrate patches. It aims to increase the proportion of patients reaching target systolic BP <140 mmHg within 1 hour of hospital admission while monitoring safety, clinical outcomes, and healthcare resource utilization.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH) is one of the most time-critical neurological emergencies. Rapid lowering of systolic blood pressure to below 140 mmHg (but not below 110 mmHg) has been associated with reduced risk of hematoma expansion and improved long-term functional outcomes. International guidelines recommend that the target blood pressure be achieved within 1 hour of hospital admission.

Traditionally, the specific class of antihypertensive agent used for acute blood pressure management in ICH was considered less important than achieving the target level. However, emerging evidence from two randomized clinical trials has raised concerns regarding the safety of transdermal long-acting nitrate patches (such as glyceryl trinitrate) in the hyperacute phase of stroke. These studies reported signals suggesting potential harm when nitrate patches were used in the early hours after symptom onset. Further, the time from derug administration to blood-pressure control is longer than intravenous administration.

In contrast, intravenous calcium channel blockers such as nicardipine have demonstrated both efficacy and safety in achieving rapid blood pressure control in acute ICH. These agents are widely used in clinical practice and are recommended in national and international guidelines.

In our institution, the standard protocol for acute blood pressure management in ICH has historically included transdermal glyceryl trinitrate patches. In light of emerging safety concerns and new recommendations, we aim to gradually implement a revised protocol centered on intravenous nicardipine. The implementation will be conducted in a cluster randomized stepwise fashion and monitored closely for its effects on blood-pressure control, safety, workflow, and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute spontaneous Intracerberal Hemorrhage confirmed by imaging
* Symptom onset to stroke center admission <24 hours
* Elevated systolic blood pressure (>140 mmHg) at admission

Exclusion Criteria:

* Secondary causes of ICH (e.g., trauma, vascular malformation)
* Presumed fatal bleeding at admission
* Short remaining life expectancy (<12 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Target blood pressure < 140 mmHg 1 hour after admission. | 1 hour after stroke center admission
  Proportion of patients reaching systolic BP <140 mmHg within 1 hour of stroke center admission

SECONDARY OUTCOMES:
Functional outcome at 3 months | 90 days (+/- 14 days)
  Proportion of patients with acceptable functional outcome at 3 months Defined as modified Rankin Scale (mRS) ≤ 3
Bed day use | 0 to 180 days
  Use of acute stroke unit bed-days
Total bed day use | 0 to 180 days
  Use of total unit bed-days (Stroke ward and in-hospital rehabilitation)
Serious adverse events | 90 days
  Proportion of patients with at least one serious adverse events (SAEs)
Hypotension | 0 to 90 days
  Proportion of patients experiencing hypotension (systolic blood rpessure <90mmHg or diastolic below 60 mmHg) during the stroke center admission
Acute kidney injury | 0 to 90 days
  Proportion of patients experiencing acute kidney injury during the stroke center admission.
  (Increase in plasma creatinine of more than 26.5 µmol/L within the past 48 hours, or Increase of 50% or more within 7 days from baseline, defined as the patient's habitual creatinine level, or Urine output of less than 0.5 mL/kg/hour over the past 6 hours despite appropriate therapy)
Reduced level of consciousness | 0 to 90 days
  Reduced level of consciousness measured as a drop of at least 2 points on the Glascow Coma Scale (range 3-15)
Intensive care unit | 0 to 90 days
  Proportion of patients admitted to the intensive carte unit
Neurosurgery | 0 to 90 days
  Incidence of surgical intervention (hematoma evacuation or external ventricular drainage) during hospital stay
Mortality | 90 days (+/- 14 days)
  All cause mortality at 90 days
Mortality | 180 days (+/- 14 days)
  All cause mortality at 180 days

OTHER OUTCOMES:
Time consumption associated with blood pressure management | From 0 to 72 hours
  Nursing time per patient related to acute blood pressure management ( Estimated via time registration in sample patients, 3-5 in each group)

IPD SHARING:
Plan to Share IPD: No
The datasets will not be shared due to legal and privacy restrictions associated with data approved for use in a quality improvement study